CLINICAL TRIAL: NCT04578626
Title: Morphological Changes in Asymptomatic Perimandibular Muscles After Dry Needling Assessed With Rehabilitative Ultrasound Imaging
Brief Title: Ultrasounds Evaluation of Asymptomatic Perimandibular Muscles Treated With Dry Needling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poliambulatorio Physio Power (Other)
Collaborators: Universidad Francisco de Vitoria (Other)
Responsible Party: Principal Investigator, Alice Botticchio, Principal investigator, Poliambulatorio Physio Power
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: US-DN-01
Record Dates: First submitted 2020-10-01; First posted 2020-10-08 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Asymptomatic State; Temporomandibular Joint; Masticatory Muscles
Keywords: ultrasonography; dry needling; physical therapy
MeSH Terms: conditions — Asymptomatic Diseases | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dry needling group (Experimental): Dry needling treatment on right or left side of the face (depending on randomization)
  Interventions: Device: dry needling
- control group (No Intervention): No treatment on left or right side of the face (depending on randomization)

INTERVENTIONS:
Device: dry needling — The use of filiform needles to stimulate muscles and connective tissues. The needle is inserted in a direction perpendicular to the skin, a local twitch response is looked for and, once found, the needle is kept in the muscle without moving for 10 seconds. No substances are injected.
  Arms: dry needling group

SUMMARY:
The articular disc of temporomandibular joint and three muscles of the cervico-facial region (temporal, masseter, sternocleidomastoid) are evaluated by means of sonographic images to observe and measure their dimensions' changes after a dry needling intervention. The participants are asymptomatic subjects and will be randomly divided in 2 groups: half of them are treated on the right side of the face, while the other half on the left side. Our hypothesis is that ultrasonography can reveal changes in the structures measured on the treated side.

DETAILED DESCRIPTION:
The trial is designed as a before-and-after study conducted on asymptomatic subjects. The aim is to assess temporomandibular joint and three perimandibular muscles (temporal, masseter, sternocleidomastoid) by means of rehabilitative ultrasound imaging, carried out by a novice clinician. These evaluations are performed before and after a dry needling treatment directed to the tree studied muscles of one side of the face. The side to be treated is randomly assigned by using a computer-generated randomization process, the other side is used as control.

One month after the treatment sonographic images are taken by the novice clinician and by an expert one. The aim is to assess the reliability of ultrasonography comparing the results of their assessments.

ELIGIBILITY:
Inclusion Criteria:

* Age major then 18 years
* Must be asymptomatic in the face/head region at the time of the visit and in the previous 6 months.

Exclusion Criteria:

* Pregnancy
* medical history of systemic disease
* current pharmacological therapy
* history of recurrent headache and/or neck pain
* presence of orofacial pain or temporomandibular symptoms assessed with the DC/TMD (Diagnostic Criteria for TemporoMandibular Disorders)
* current use of a bite during sleep

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
mean of temporomandibular joint disc thickness | Baseline (before the treatment), immediately after the treatment, one month after the treatment
  the distance between the opposing surfaces of the disc (cm)
mean of temporal muscle thickness | Baseline (before the treatment), immediately after the treatment, one month after the treatment
  the distance between the opposing borders of the muscle, along the transverse axis of the muscle (cm)
mean of masseter muscle thickness | Baseline (before the treatment), immediately after the treatment, one month after the treatment
  the distance between the superficial and the deep border of the muscle (cm)
mean of masseter muscle width | Baseline (before the treatment), immediately after the treatment, one month after the treatment
  the distance between the opposing extremities of the muscle along the transverse axis of the muscle (cm)
mean of masseter muscle cross-sectional area | Baseline (before the treatment), immediately after the treatment, one month after the treatment
  the area of the muscle in transversal plan measured after drawing the outline of the muscle in an image obtained with the panoramic view function (cm2)
mean of sternocleidomastoid muscle thickness | Baseline (before the treatment), immediately after the treatment, one month after the treatment
  the distance between the superficial and the deep border of the muscle (cm)
mean of sternocleidomastoid muscle width | Baseline (before the treatment), immediately after the treatment, one month after the treatment
  the distance between the opposing extremities of the muscle along the transverse axis of the muscle (cm)
mean of sternocleidomastoid muscle cross-sectional area | Baseline (before the treatment), immediately after the treatment, one month after the treatment
  the area of the muscle in transversal plan measured after drawing the outline of the muscle in an image obtained with the panoramic view function (cm2)

SECONDARY OUTCOMES:
mean of maximum mouth opening | Baseline (before the treatment), one month after the treatment
  the distance between the superior border of inferior front teeth and the inferior border of superior front teeth (cm)

CONTACTS AND LOCATIONS:
Overall Officials: Alice Botticchio, PT, OMPT, Principal Investigator — Poliambulatorio PhysioPower, Brescia, Italy
Locations (1):
- Universidad Francisco de Vitoria, Pozuelo de Alarcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
We are not intentioned to share the participant data as our outcomes are subjectively evaluated by the use of ultrasonography. We don't believe it will be helpful for other researches as the results will be interpreted by our assessors.

REFERENCES:
- [Background] Schiffman E, Ohrbach R, Truelove E, Look J, Anderson G, Goulet JP, List T, Svensson P, Gonzalez Y, Lobbezoo F, Michelotti A, Brooks SL, Ceusters W, Drangsholt M, Ettlin D, Gaul C, Goldberg LJ, Haythornthwaite JA, Hollender L, Jensen R, John MT, De Laat A, de Leeuw R, Maixner W, van der Meulen M, Murray GM, Nixdorf DR, Palla S, Petersson A, Pionchon P, Smith B, Visscher CM, Zakrzewska J, Dworkin SF; International RDC/TMD Consortium Network, International association for Dental Research; Orofacial Pain Special Interest Group, International Association for the Study of Pain. Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) for Clinical and Research Applications: recommendations of the International RDC/TMD Consortium Network* and Orofacial Pain Special Interest Groupdagger. J Oral Facial Pain Headache. 2014 Winter;28(1):6-27. doi: 10.11607/jop.1151. PMID 24482784
- [Background] de-Pedro-Herraez M, Mesa-Jimenez J, Fernandez-de-Las-Penas C, de-la-Hoz-Aizpurua JL. Myogenic temporomandibular disorders: Clinical systemic comorbidities in a female population sample. Med Oral Patol Oral Cir Bucal. 2016 Nov 1;21(6):e784-792. doi: 10.4317/medoral.21249. PMID 27694784
- [Background] Ries LG, Alves MC, Berzin F. Asymmetric activation of temporalis, masseter, and sternocleidomastoid muscles in temporomandibular disorder patients. Cranio. 2008 Jan;26(1):59-64. doi: 10.1179/crn.2008.008. PMID 18290526
- [Background] Dahlstrom L, Carlsson GE. Temporomandibular disorders and oral health-related quality of life. A systematic review. Acta Odontol Scand. 2010 Mar;68(2):80-5. doi: 10.3109/00016350903431118. PMID 20141363
- [Background] Oliveira LK, Almeida Gde A, Lelis ER, Tavares M, Fernandes Neto AJ. Temporomandibular disorder and anxiety, quality of sleep, and quality of life in nursing professionals. Braz Oral Res. 2015;29:S1806-83242015000100265. doi: 10.1590/1807-3107BOR-2015.vol29.0070. PMID 26039910
- [Background] Weiss RC, Oostrom-Ram T. Inhibitory effects of ribavirin alone or combined with human alpha interferon on feline infectious peritonitis virus replication in vitro. Vet Microbiol. 1989 Jul;20(3):255-65. doi: 10.1016/0378-1135(89)90049-7. PMID 2549687
- [Background] Emshoff R, Bertram S, Strobl H. Ultrasonographic cross-sectional characteristics of muscles of the head and neck. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 1999 Jan;87(1):93-106. doi: 10.1016/s1079-2104(99)70302-1. PMID 9927088
- [Background] Djordjevic O, Djordjevic A, Konstantinovic L. Interrater and intrarater reliability of transverse abdominal and lumbar multifidus muscle thickness in subjects with and without low back pain. J Orthop Sports Phys Ther. 2014 Dec;44(12):979-88. doi: 10.2519/jospt.2014.5141. Epub 2014 Nov 3. PMID 25366083
- [Background] Strini PJ, Strini PJ, Barbosa Tde S, Gaviao MB. Assessment of thickness and function of masticatory and cervical muscles in adults with and without temporomandibular disorders. Arch Oral Biol. 2013 Sep;58(9):1100-8. doi: 10.1016/j.archoralbio.2013.04.006. Epub 2013 May 16. PMID 23684155
- [Background] Pallegama RW, Ranasinghe AW, Weerasinghe VS, Sitheeque MA. Influence of masticatory muscle pain on electromyographic activities of cervical muscles in patients with myogenous temporomandibular disorders. J Oral Rehabil. 2004 May;31(5):423-9. doi: 10.1111/j.1365-2842.2004.01266.x. PMID 15140167
- [Background] Fedorowicz Z, van Zuuren EJ, Schoones J. Botulinum toxin for masseter hypertrophy. Cochrane Database Syst Rev. 2013 Sep 9;2013(9):CD007510. doi: 10.1002/14651858.CD007510.pub3. PMID 24018587
- [Background] Ariji Y, Sakuma S, Izumi M, Sasaki J, Kurita K, Ogi N, Nojiri M, Nakagawa M, Takenaka M, Katsuse S, Ariji E. Ultrasonographic features of the masseter muscle in female patients with temporomandibular disorder associated with myofascial pain. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2004 Sep;98(3):337-41. doi: 10.1016/j.tripleo.2004.06.068. PMID 15356473
- [Background] Gonzalez-Perez LM, Infante-Cossio P, Granados-Nunez M, Urresti-Lopez FJ, Lopez-Martos R, Ruiz-Canela-Mendez P. Deep dry needling of trigger points located in the lateral pterygoid muscle: Efficacy and safety of treatment for management of myofascial pain and temporomandibular dysfunction. Med Oral Patol Oral Cir Bucal. 2015 May 1;20(3):e326-33. doi: 10.4317/medoral.20384. PMID 25662558
- [Background] Dunning J, Butts R, Mourad F, Young I, Flannagan S, Perreault T. Dry needling: a literature review with implications for clinical practice guidelines. Phys Ther Rev. 2014 Aug;19(4):252-265. doi: 10.1179/108331913X13844245102034. PMID 25143704
- [Background] Diracoglu D, Vural M, Karan A, Aksoy C. Effectiveness of dry needling for the treatment of temporomandibular myofascial pain: a double-blind, randomized, placebo controlled study. J Back Musculoskelet Rehabil. 2012;25(4):285-90. doi: 10.3233/BMR-2012-0338. PMID 23220812
- [Background] Turo D, Otto P, Hossain M, Gebreab T, Armstrong K, Rosenberger WF, Shao H, Shah JP, Gerber LH, Sikdar S. Novel Use of Ultrasound Elastography to Quantify Muscle Tissue Changes After Dry Needling of Myofascial Trigger Points in Patients With Chronic Myofascial Pain. J Ultrasound Med. 2015 Dec;34(12):2149-61. doi: 10.7863/ultra.14.08033. Epub 2015 Oct 21. PMID 26491094
- [Background] Emshoff R, Bertram S, Rudisch A, Gassner R. The diagnostic value of ultrasonography to determine the temporomandibular joint disk position. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 1997 Dec;84(6):688-96. doi: 10.1016/s1079-2104(97)90374-7. PMID 9431541
- [Background] Raadsheer MC, Van Eijden TM, Van Spronsen PH, Van Ginkel FC, Kiliaridis S, Prahl-Andersen B. A comparison of human masseter muscle thickness measured by ultrasonography and magnetic resonance imaging. Arch Oral Biol. 1994 Dec;39(12):1079-84. doi: 10.1016/0003-9969(94)90061-2. PMID 7717890
- [Background] Cagnie B, Dewitte V, Barbe T, Timmermans F, Delrue N, Meeus M. Physiologic effects of dry needling. Curr Pain Headache Rep. 2013 Aug;17(8):348. doi: 10.1007/s11916-013-0348-5. PMID 23801002
- [Background] Smith P, Mosscrop D, Davies S, Sloan P, Al-Ani Z. The efficacy of acupuncture in the treatment of temporomandibular joint myofascial pain: a randomised controlled trial. J Dent. 2007 Mar;35(3):259-67. doi: 10.1016/j.jdent.2006.09.004. Epub 2006 Nov 13. PMID 17095133
- [Background] Hides J, Richardson C, Jull G, Davies S. Ultrasound imaging in rehabilitation. Aust J Physiother. 1995;41(3):187-93. doi: 10.1016/S0004-9514(14)60429-3. PMID 25026042
- [Background] Hodges PW. Ultrasound imaging in rehabilitation: just a fad? J Orthop Sports Phys Ther. 2005 Jun;35(6):333-7. doi: 10.2519/jospt.2005.0106. No abstract available. PMID 16001904
- [Background] Teyhen DS. Rehabilitative ultrasound imaging for assessment and treatment of musculoskeletal conditions. Man Ther. 2011 Feb;16(1):44-5. doi: 10.1016/j.math.2010.06.012. Epub 2010 Aug 1. No abstract available. PMID 20678956
- [Background] Bubnov RV. The use of trigger point "dry" needling under ultrasound guidance for the treatment of myofascial pain (technological innovation and literature review). Lik Sprava. 2010 Jul-Sep;(5-6):56-64. PMID 21485754